CLINICAL TRIAL: NCT04400760
Title: The Effect of Dapagliflozin on Platelet Function testinG Profiles in Diabetic PatiEnts: The EDGE Study.
Brief Title: The Effect of Dapagliflozin on Platelet Function testinG Profiles in Diabetic PatiEnts.
Acronym: EDGE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Naveen Seecheran, Principal Investigator, The University of The West Indies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC-SA.0284/03/2020
Record Dates: First submitted 2020-05-19; First posted 2020-05-26 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Platelet Dysfunction
Keywords: dapagliflozin; SGLT2i

STUDY DESIGN:
Intervention Model Description: The study will be of a prospective, open-label trial design over a 2-year period. Patients at the Eric Williams Medical Sciences Complex (EWMSC), Mt. Hope, Trinidad and Tobago will be screened for potential eligibility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- DAPA Tx (Other): This arm will comprise the participants who are administered Dapagliflozin 10mg per oral once daily for 2 weeks.
  Interventions: Drug: DAPA Tx

INTERVENTIONS:
Drug: DAPA Tx — The intervention, dapagliflozin will be administered 10mg per oral daily for two weeks.

SUMMARY:
Sodium GLucose Transport 2 inhibitors (SGLT2I), including dapagliflozin, reduce the likelihood of hospitalization for heart failure and death in persons with type 2 diabetes, of which the mechanism has not been fully elucidated. The mechanistic effects of dapagliflozin on platelet function profiles have not yet been ascertained. It remains unclear if this reduction in cardiovascular death is mediated by decreased platelet reactivity.

DETAILED DESCRIPTION:
Diabetes is highly prevalent in our setting. Dapagliflozin is now considered first-line treatment for diabetes, especially in the cardiovascular arena. The standard prescribed dosages of dapagliflozin will be employed in the research study (5 or 10 mg once daily). The reason the study team is interested in performing this study in our local setting is that if dapagliflozin does show a beneficial effect with either diabetic control or an antiplatelet effect, the team can then inform the Ministry of Health to acquire these relatively expensive medications in place of the older, less effective anti-diabetic drugs. The team has to demonstrate that they work effectively and safely in our population before approaching regulatory bodies with a robust recommendation that they are made available in the public healthcare sector. The patients that are to be selected will be relatively controlled on their current regimen, and thus not "miss out" on these medications after the study has been concluded as they are all available on the chronic disease assistance program (CDAP) such as metformin, gliclazide and insulin therapies. The study will aim to determine if dapagliflozin does demonstrate other latent antiplatelet effects that can potentially affect the cardiovascular/hematologic systems that have not investigated before.

ELIGIBILITY:
Inclusion Criteria:

1. between 18 and 74 years of age,
2. have stable coronary artery disease and diabetes mellitus, already on DAPT with aspirin and clopidogrel for at least 6 months,
3. not on any physician-prescribed medications or complementary/alternative therapies.

Exclusion Criteria:

1. presence of active internal bleeding or history of bleeding diathesis or clinical findings associated with an increased risk of bleeding,
2. history of ischemic or hemorrhagic stroke, transient ischemic attack, intracranial neoplasm, arteriovenous malformation, or aneurysm,
3. history of clinical and/or hemodynamic instability,
4. within 1 month of placement of a bare-metal stent,
5. within 30 days of coronary artery bypass graft surgery or PCI without a stent placed,
6. planned coronary revascularization,
7. treatment with fibrin-specific fibrinolytic therapy <24 h or non-fibrin-specific fibrinolytic therapy <48 h,
8. use of an oral anticoagulation agent or international normalized ratio >1.5,
9. body weight <60 kg,
10. age >75 years,
11. hemoglobin <10 g/dL,
12. platelet count <100×106/μL,
13. creatinine >2 mg/dL,
14. hepatic enzymes >2.5 times the upper limit of normal,
15. pregnancy and/or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naveen A Seecheran, MBBS MSc, Principal Investigator — The University of The West Indies
Locations (1):
- Eric Williams Medical Sciences Complex, Port of Spain, North Central, Trinidad and Tobago

REFERENCES:
- [Derived] Seecheran N, Grimaldos K, Ali K, Grimaldos G, Richard S, Ishmael A, Gomes C, Karan A, Seecheran R, Seecheran V, Persad S, Abdullah H, Peram L, Dookeeram D, Giddings S, Motilal S, Raza S, Tello-Montoliu A, Schneider D. The Effect of Dapagliflozin on Platelet Function Testing Profiles in Diabetic Patients: The EDGE Pilot Study. Cardiol Ther. 2021 Dec;10(2):561-568. doi: 10.1007/s40119-021-00242-6. Epub 2021 Oct 13. PMID 34643895

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DAPA Tx
Started | 40
Completed | 27
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | DAPA Tx
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 0
  More than one race | 3
  Unknown or Not Reported | 0
PRU [Mean (Standard Deviation); unit: PRU] | 160.93 (1)

OUTCOME MEASURES:

1. Primary Outcome: Platelet Reactions Units Pre-DAPA Tx and Post-DAPA Tx
Description: Platelet Reaction units at baseline and post-DAPA Tx treatment with dapagliflozin
Time Frame: Baseline (0 weeks) to Completion (2 weeks) after Dapagliflozin
Measure: Mean (95% Confidence Interval); unit: PRU
Arm/Group | DAPA Tx
Number analyzed (Participants) | 27
PRU | 160.93 [129.28 to 192.57]

ADVERSE EVENTS:
Time Frame: 28 days.
Arm/Group | DAPA Tx
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT04400760/Prot_SAP_001.pdf